CLINICAL TRIAL: NCT04879147
Title: Observational and Diagnostical Study on Transient Allostatic Responses of Thyroid Function After Syncopation and Seizure (Thyro-Syncope)
Brief Title: Observational and Diagnostical Study on Transient Allostatic Responses of Thyroid Function After Syncopation and Seizure
Acronym: Thyro-Syncope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Bergmannsheil University Hospitals (Unknown)
Responsible Party: Principal Investigator, PD Dr. Johannes W. Dietrich, MD, Consultant Endocrinologist, Ruhr University of Bochum
Other Study IDs: 21-7171; DRKS00025266 (Registry Identifier: DRKS)
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Syncope; Seizures
Keywords: thyroid allostasis; TACITUS; syncope; seizure; loss of consciousness
MeSH Terms: conditions — Syncope; Seizures; Unconsciousness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum specimens are stored as aliquots at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Syncope: Subjects admitted immediately after syncopation.
  Interventions: Diagnostic Test: Evalution of thyroid function
- Seizre: Subject admitted immediately after cerebarl seizure
  Interventions: Diagnostic Test: Evalution of thyroid function

INTERVENTIONS:
Diagnostic Test: Evalution of thyroid function — Determination of TSH, free T4, free T3, SPINA-GT, SPINA-GD and Jostel's TSH index

SUMMARY:
Changes of thyroid function may occur after short loss of consciousness, but they haven't been systematically evaluated up to now, although occasional observations suggest temporal increases in TSH concentration.

This study aims at assessing transient changes of biomarkers of thyroid function after syncopation and seizure.

Results of the study might contribute to an improved detection rate of thyrotoxicosis.

DETAILED DESCRIPTION:
Transient allostatic responses of thyroid function have been described in critical illness. Own observations suggest similar reactive responses after syncopation and cerebral seizures. They are marked especially by increased concentration of serum thyrotropin (TSH), suggesting a type 2 allostatic response. However, changes of thyroid function after temporal loss of consciousness haven't been systematically evaluated up to now. Current diagnostic guidelines recommend primarily the determination of serum TSH concentration for screening of thyroid function, and the measurement of peripheral thyroid hormones (T4 and/or T3) is only recommended if TSH determination results in pathological values. This TSH reflex strategy may be misleading after short-term loss of consciousness.

This study aims at assessing the prevalence of allostatic responses of thyroid function after events of syncopation or seizure and at investigating the consecutive temporal development of biomarkers of thyroid function. An additional aim includes the diagnostic value of TSH determination, compared to measurement of free thyroid hormones, for thyroid dysfunction after syncopation or seizure.

Results of this study might contribute to an improved detection rate of thyrotoxicosis. In cases of medical emergencies and in-patient treatment interventions with a significant iodine load are common, including the application of iodinated radiocontrast agents and amiodarone. In this setting, undetected hyperthyroidism may lead to thyroid storm, which is associated with a high mortality.

ELIGIBILITY:
Inclusion Criteria:

* Admission after syncope or seizure
* Age of 18 years or older
* First bleed not later than two hours after event (syncope or seizure)
* Written informed consent obtained

Exclusion Criteria:

* Results of thyroid hormones not available within two hours after event
* Pituitary dysfunction
* Thyroid dysfunction
* Use of iodinated radiocontrast agents less than three months ago
* Therapy with amiodarone in the previous three years
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible are subjects addmitted for in-patient treatment after syncope or cerebral seicure
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
Prevalence of allostatic responses of thyroid function after short-term loss of consciousness | 2 hours
  Prevalence of increased TSH immediately after syncope or seizure

SECONDARY OUTCOMES:
Time series of thyroid function after short-term loss of consciousness | 72 hours
  Temporal evolution of TSH and thyroid hormone concentration during three days after syncope or seicure
Diagnostic value of TSH after short-term loss of consciousness | 72 hours
  Sensitivity, specificitay and likelihood ratios of TSH compared to free T4 and free T3 after syncopation or seizure

CONTACTS AND LOCATIONS:
Overall Officials: Johannes W Dietrich, M.D., Principal Investigator — Bergmannsheil University Hospitals
Locations (4):
- Germany (4):
  - Institute of Clinical Chemistry, Transfusion and Laboratory Medicine, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia
  - Medical Hospital I, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia
  - Medical Hospital II, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia
  - Neurological University Hospital and Clinics, Bergmannsheil University Hospitals, Ruhr University of Bochum, Bochum, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared upon request.

REFERENCES:
- [Background] Aweimer A, El-Battrawy I, Akin I, Borggrefe M, Mugge A, Patsalis PC, Urban A, Kummer M, Vasileva S, Stachon A, Hering S, Dietrich JW. Abnormal thyroid function is common in takotsubo syndrome and depends on two distinct mechanisms: results of a multicentre observational study. J Intern Med. 2021 May;289(5):675-687. doi: 10.1111/joim.13189. Epub 2020 Nov 12. PMID 33179374
- [Background] Chatzitomaris A, Hoermann R, Midgley JE, Hering S, Urban A, Dietrich B, Abood A, Klein HH, Dietrich JW. Thyroid Allostasis-Adaptive Responses of Thyrotropic Feedback Control to Conditions of Strain, Stress, and Developmental Programming. Front Endocrinol (Lausanne). 2017 Jul 20;8:163. doi: 10.3389/fendo.2017.00163. eCollection 2017. PMID 28775711
- [Background] Dietrich JW, Stachon A, Antic B, Klein HH, Hering S. The AQUA-FONTIS study: protocol of a multidisciplinary, cross-sectional and prospective longitudinal study for developing standardized diagnostics and classification of non-thyroidal illness syndrome. BMC Endocr Disord. 2008 Oct 13;8:13. doi: 10.1186/1472-6823-8-13. PMID 18851740
- [Background] Dietrich JW, Muller P, Schiedat F, Schlomicher M, Strauch J, Chatzitomaris A, Klein HH, Mugge A, Kohrle J, Rijntjes E, Lehmphul I. Nonthyroidal Illness Syndrome in Cardiac Illness Involves Elevated Concentrations of 3,5-Diiodothyronine and Correlates with Atrial Remodeling. Eur Thyroid J. 2015 Jun;4(2):129-37. doi: 10.1159/000381543. Epub 2015 May 23. PMID 26279999
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554
- [Background] Dietrich JW, Hoermann R, Midgley JEM, Bergen F, Muller P. The Two Faces of Janus: Why Thyrotropin as a Cardiovascular Risk Factor May Be an Ambiguous Target. Front Endocrinol (Lausanne). 2020 Oct 26;11:542710. doi: 10.3389/fendo.2020.542710. eCollection 2020. PMID 33193077
- [Background] Fitzgerald SP, Bean NG, Falhammar H, Tuke J. Clinical Parameters Are More Likely to Be Associated with Thyroid Hormone Levels than with Thyrotropin Levels: A Systematic Review and Meta-Analysis. Thyroid. 2020 Dec;30(12):1695-1709. doi: 10.1089/thy.2019.0535. Epub 2020 Jun 4. PMID 32349628
- [Background] Goldstein DS. Adrenal responses to stress. Cell Mol Neurobiol. 2010 Nov;30(8):1433-40. doi: 10.1007/s10571-010-9606-9. PMID 21061156
- [Background] Stanculescu D, Larsson L, Bergquist J. Hypothesis: Mechanisms That Prevent Recovery in Prolonged ICU Patients Also Underlie Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). Front Med (Lausanne). 2021 Jan 28;8:628029. doi: 10.3389/fmed.2021.628029. eCollection 2021. PMID 33585528